CLINICAL TRIAL: NCT04174417
Title: Effect of Hypotensive Anesthesia on Cerebral Perfusion and Blood Antioxidant Levels and HIF 1a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Ayşe ŞENCAN, MD, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Ayse01
Record Dates: First submitted 2019-11-12; First posted 2019-11-22 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Hypoxemia During Surgery; Hypoxia, Brain
Keywords: hypotensive anesthesia; HIF 1a; Brain Hypoxia; tissue hypoxia
MeSH Terms: conditions — Hypoxia, Brain | interventions — Blood Pressure; Arterial Pressure

STUDY DESIGN:
Intervention Model Description: A total of 60 ASA 1-2 patients aged between 18-75 who underwent elective rhinoplasty and orthognathic surgery were included the study.The patients were divided into two groups. One group received hypotensive anesthesia according to MBP an done group received SBP. Continuous regional cerebral oxygen saturation was monitored by NIRS in both groups. Blood samples were taken from all patients before anesthesia induction and at the and of the operation and stored for TAS, TOS, HIF 1a. At the and of the operation patients were fallowed in the post anesthesia care unit for 30 minutes and pain and nause vomiting scores were evaluated. İn addition, surgical satisfaction and bleeding scores and anesthetic consumption of both groups were recorded
Who Masked: Participant
Masking Description: The investigators diveded the patients to two groups. Patients were divided into two groups with a lottery. Surgeons did not know which hypotensive anesthesia technique were used. And surgeons evaluated surgical satisfaction and bleeding scores
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systolic blood pressure (SBP) (Active Comparator): Systolic blood pressure (SBP) for group 1 patients 80-90 mmHg
  Interventions: Procedure: systolic blood pressure (SBP)
- mean blood pressure (MBP) (Active Comparator): Mean blood pressure (MBP) for group 2 patients 50-65 mmHg
  Interventions: Procedure: mean blood pressure (MBP)

INTERVENTIONS:
Procedure: systolic blood pressure (SBP) — Systolic blood pressure (SBP) 80-90 mmHg remifentanil infusion was applied to Group 1 patients. In addition to remifentanil infusion, 0.002 μg.kg of glycerol trinitrate (Perlinganit) was administered as an intermittent bolus in patients who needed to achieve target blood pressure. All patients received 5-8 ml / kg / h IV infusion of balanced electrolyte solution (Isolyte-S) during the operation.
  Hemodynamic parameters (HR, SBP, OCD), BIS, SpO2 and NIRS were recorded at 5 minute intervals. At the end of the operation, 3 ml of blood was taken from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory
  Arms: systolic blood pressure (SBP)
Procedure: mean blood pressure (MBP) — For group 2, remifentanil infusion was performed with a mean blood pressure (OCD) of 50-65 mmHg. In addition to remifentanil infusion, 0.002 μg.kg of glycerol trinitrate (Perlinganit) was administered as an intermittent bolus in patients who needed to achieve target blood pressure. All patients received 5-8 ml / kg / h IV infusion of balanced electrolyte solution (Isolyte-S) during the operation.
  Hemodynamic parameters (HR, SBP, OCD), BIS, SpO2 and NIRS were recorded at 5 minute intervals. At the end of the operation, 3 ml of blood was taken from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory.
  Arms: mean blood pressure (MBP)

SUMMARY:
The aim of this study to evaluate the patients who underwent controlled hypotensive anesthesia under standardized depth of anesthesia; preoperative and postoperative blood HIF 1a, TAS, TOS measurement and cerebral perfusion evaluation with NIRS and to investigate tissue hypoxia secondary to hypotensive anesthesia and the changes of the mediators at the tissue level and which blood pressure parameters are related.

DETAILED DESCRIPTION:
Controlled hypotension is the voluntary reversible reduction of arterial blood pressure. Hypotensive anesthesia is a method of anesthesia in which blood pressure is reduced in a controlled manner, especially in certain surgeries. İt reduces intraoperative bleeding and need for blood transfusion and provides a clean surgical vision in narrow-field surgeries or with high bleeding potential. Hypotensive anesthesia can be performed according to mean blood pressure (MBP) or systolic blood pressure (SBP).

A non-invasive cerebral oximeter is used to see the changes in the brain due to high oxygen-dependent metabolism during induction and maintenance of anesthesia.

Hypoxia inducible factor (HIF) is a transcription factor involved in cell adaptation mechanism activated in response to hypoxia.

The biological activity of HIF 1 is determined by the expression and activity of the HIF 1a subunit.

Total antioxidant status (TAS) shows the total effect of all antioxidants in the human body and total oxidant status (TOS) shows the total effect of oxidants.

Near Infrared Spectroscopy (NIRS) allows continuous and non-invasive monitoring of cerebral oxygenation. HIF 1a, TAS and TOS are laboratory markers that predict tissue oxygenation and perfusion.

Hypotensive anesthesia can be performed according to both MBP and SBP. However, in our study that follow-up MBP is more advantageous/protective, although it is not supported by very strong data. The investigators recommend hypotensive anesthesia compared to MBP; but further studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* ASA Physical Status Classification System 1-2
* Undergoing to Elective rhinoplasty or maxillofacial surgery

Exclusion Criteria:

* 1. Those with SVO history 2. Patients with carotid stenosis and cardiac failure 3. Chronic smoking 4. Patients with allergies to drugs to be used 5. Patients without intraoperative hypotension 6. Presence of morbid obesity (BMI> 40 kg / m2) 7. Patients who refused to participate in the study

Termination criteria

1. Development of severe hypotension and bradycardia during measurements
2. Development of severe drug allergy during follow-up
3. In the event of any complications related to the surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the relationship between hypotensive anesthesia technique and brain hypoxia by the rate of NIRS | intraoperative 2 hours
  The investigators used to detect brain hypoxia with Near Infrared Spectroscopy (NIRS) (INVOS 5100 Medtronic).
  Near Infrared measurement, primary absorbing molecules in tissue are metal complex chromophores such as hemoglobin, bilirubin and cytochrome.
  The absorption spectra of deoxyhemoglobin (Hb) range between 650-1000 nm, the oxyhemoglobin (Hb02) absorption spectra range between 700-1150 and the cytochrome oxidase aa3 (Caa3) absorption spectra range from 820-840 nm.
  NIRS measures the ratio of oxyhemoglobin to total hemoglobin at a depth of 2.5-3 cm in the area under the sensor.This ratio represents regional cerebral oxygen (RsO2) saturation.
  RSO2 below 40% or more than 25% decrease in baseline is associated with neurological dysfunction and side effects. A 15-20% reduction or less than 50% of the baseline is considered a critical threshold and requires action.
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by HIF1a | Change from Baseline HIF 1a at 2 hours
  Under normoxic conditions, HIF 1a protein can hardly be detected, but when hypoxia starts, its expression starts within 2 minutes and peaks at 4-8 hours of hypoxia.
  3 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia induction for measure HIF 1a,TAS and TOS. At the end of the operation, 3 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by the concentration of TAS | Change from Baseline TAS levels at 2 hours
  Plasma TAS and TOS levels are measured with a commercial kit developed by Erel. Values for plasma TAS are expressed in millimeters by the Trolox value per liter.
  3 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia induction for measure HIF 1a,TAS and TOS. At the end of the operation, 3 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.
Evaluation of the relationship between hypotensive anesthesia technique and tissue hypoxia by the concentration of TOS | Change from Baseline TOS levels at 2 hours
  Measurement for TOS is calibrated with hydrogen peroxide and the results are expressed in micromolar by the hydrogen peroxide value per liter (mmol H2O2 equiv / L).
  3 ml blood was taken into MiniCollect® tubes from the venous cannula placed before anesthesia induction for measure HIF 1a,TAS and TOS. At the end of the operation, 3 ml of blood was taken again from the untreated arm of all patients to the HIF1a, TAS and TOS values and sent to the biochemistry laboratory. The collected blood was centrifuged at 2000 x g for 10 minutes and the separated sera were sent to the biochemical laboratory to be stored at -80 ° C until the study was performed.

SECONDARY OUTCOMES:
surgical satisfaction | postoperative 1 minute
  At the end of the surgery surgeons evaluated surgical satisfaction. the investigators used surgeon satisfaction score which one is performing like that 1- bad 2-moderate 3-good 4-excellent
bleeding scores | postoperative 1 minute
  At the end of the surgery surgeons evaluated bleeding scores. the investigators used bleeding score which one is performing like that 0-No bleeding 1-minor bleeding no aspiration required 2- Minor bleeding, aspiration required 3-minor bleeding, frequent aspiration required, 4-Moderate bleeding, visible only with aspiration 5- Severe bleeding, frequent aspiration required and very hard to perform surgery
anesthetic consumption | postoperative 1 minute
  Standard anesthesia induction and propofol and remifentanil infusion were applied to all patients with TIVA technique.

CONTACTS AND LOCATIONS:
Overall Officials: Hayrettin Daşkaya, MD, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No